CLINICAL TRIAL: NCT06293339
Title: Durability of Protection After Single Immunisation With Genetically Attenuated Plasmodium Falciparum ∆mei2 (GA2) Sporozoites - a Follow-up, Controlled Human Malaria Rechallenge Study
Brief Title: Durability of Protection After Single Immunisation With GA2 Sporozoites (CoGA-Rechallenge)
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, Meta Roestenberg, Prof, Leiden University Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CoGA-Re
Record Dates: First submitted 2024-02-27; First posted 2024-03-05 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Malaria,Falciparum
MeSH Terms: conditions — Malaria, Falciparum | interventions — 1-acetyl-1,2,3,3a,8,8a-hexahydro-8a-hydroxy-5-methoxypyrrolo(2,3-b)indole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rechallenge group (Experimental): Previous CoGA phase 1 study participants who were immunised with GA2 and who did not develop blood-stage malaria during CHMI (protected)
  Interventions: Biological: CHMI with 3D7 malaria
- Infection control group (Placebo Comparator): Malaria-naïve participants who have not been previously vaccinated with GA2
  Interventions: Biological: CHMI with 3D7 malaria

INTERVENTIONS:
Biological: CHMI with 3D7 malaria — Controlled human malaria infection with 3D7 malaria through mosquito bites

SUMMARY:
This study will assess the durability of protection of a single immunisation with the Genetically Attenuated Parasite 2 (GA2) against controlled human malaria infection by rechallenging previously immunised and protected participants from the CoGA study (NCT05468606)

DETAILED DESCRIPTION:
This will be a non-randomised, open-label, controlled human malaria infection study that will consist of two study arms: the rechallenge group and infection controls. The rechallenge group consists of study participants from the CoGA study (phase I) who received single immunisation with GA2 and were protected during subsequent CHMI, while infection controls are newly recruited, malaria-naïve study participants. All participants will undergo CHMI through the bites of 5 mosquitos infected with wild-type 3D7 sporozoites. From day 6 to 21 after CHMI, participants will be followed daily on an out-patient basis to determine parasite loads detected by a quantitative polymerase chain reaction (qPCR). As soon as parasitaemia is detected (cut-off >100p/mL), or at the latest 28 days after CHMI, participants will be treated with a curative regimen of antimalarials.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is aged ≥18 and ≤35 years and in good health.
2. Rechallenge group only: participation in CoGA study, having received immunisation with 1x 50 GA2-infected MB, and protected during subsequent CHMI.
3. Participant has adequate understanding of the procedures of the study and agrees to abide strictly thereby.
4. Participant is able to communicate well with the investigator.
5. Participant is available to attend all essential study visits.
6. Participant agrees that his/her general practitioner (GP) will be informed about participation in the study.
7. Participant agrees to refrain from blood donation to Sanquin or for other purposes. throughout the study period and for a defined period thereafter according to Sanquin guidelines.
8. Participants of child bearing potential (i.e., have an uterus and are neither surgically sterilized nor post-menopausal) agree to use adequate contraception and to not breastfeed for the duration of study.
9. Participant agrees to refrain from intensive physical exercise (disproportionate to the participants' usual daily activity or exercise routine) for twenty-one days following the immunization and during the malaria challenge period.
10. Participant signs informed consent.

Exclusion Criteria:

1. Any history, or evidence at screening, of clinically significant symptoms, physical signs or abnormal laboratory values suggestive of systemic conditions which could compromise the health of the participant during the study or interfere with the interpretation of the study results. These include, but are not limited to, any of the following:

   a. Body Mass Index (BMI) >35.0 kg/m2 at screening. b. An elevated risk of cardiovascular disease, defined as: i. An estimated ten-year risk of fatal cardiovascular disease of ≥5% at screening, as determined by the Systematic Coronary Risk Evaluation 2 (SCORE2) .

   ii. History, or evidence at screening, of clinically significant arrhythmia's, prolonged QT-interval or other clinically relevant ECG abnormalities; or iii. A positive family history of cardiac events in first- or second-degree relatives (according to the system used in medical genetics) <50 years old.

   b. Known functional asplenia, sickle cell trait/disease, thalassemia trait/disease or G6PD deficiency.

   c. History of epilepsy in the period of five years prior to study onset, even if no longer on medication.

   d. Positive HIV, HBV or HCV screening tests. e. Chronic use of i) immunosuppressive drugs, ii) antibiotics, iii) or other drugs that might have an influence on the immune system (excluding inhaled and topical corticosteroids and incidental use of oral anti-histamines), within three months prior to study onset or expected use of such during the study period.

   f. Skin disease affecting the site of administration in such a way that administration of mosquito bites is deemed impossible by investigator.

   g. History of malignancy of any organ system (other than localized basal cell carcinoma of the skin), treated or untreated, within the past five years.

   h. Any history of treatment for severe psychiatric disease by a psychiatrist in the past year.

   i. History of drug or alcohol abuse interfering with normal social functioning in the period of one year prior to study onset, positive urine toxicology test for cocaine or amphetamines at screening.
2. For participants of child bearing potential: breastfeeding, or positive serum pregnancy test prior to CHMI.
3. Infection controls only: any history of malaria or previous participation in any malaria (vaccine) study or CHMI.
4. Known hypersensitivity to or contra-indications for both atovaquone/proguanil or artemether/lumefantrine. QT prolonging drugs are only considered an exclusion criterion when QT prolongation is observed at the ECG at screening.
5. A history of severe (allergic) reactions to mosquito bites.
6. Participation in any other clinical study assessing an investigational medical product in the 30 days prior to the start of the study or during the study period.
7. Any condition or situation that could influence the independent consent of participant (e.g. being a direct colleague or family member of study personnel).
8. Any other condition or situation that would, in the opinion of the investigator, place the participant at an unacceptable risk of injury or render the participant unable to meet the requirements of the protocol or would compromise the integrity of the data.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Protective efficacy | Moment of CHMI to antimalarial treatment (28 days post CHMI)
  Proportion of participants that do not develop parasitaemia (qPCR >100p/mL) (sterile protection) after CHMI (re)challenge in participants with prior, single GA2 immunisation compared to infection controls.
Time to parasitaemia | Moment of CHMI to antimalarial treatment (28 days post CHMI)
  The time to parasitaemia (qPCR >100 p/mL) (prepatent period) after CHMI (re)challenge between participants with prior, single GA2 immunisation and infection controls.

SECONDARY OUTCOMES:
Humoral immune responses after homologous CHMI rechallenge | Moment of CHMI up to182 days post CHMI
  Difference in concentration of anti-CSP antibodies between groups as assessed by ELISA.
Cellular immune responses after homologous CHMI rechallenge | Moment of CHMI up to182 days post CHMI
  Difference in percentage of CD4+ and CD8+ T-cells producing IFN-γ between groups as assessed by flow cytometry

CONTACTS AND LOCATIONS:
Overall Officials: Meta Roestenberg, Prof, Principal Investigator — LUMC

IPD SHARING:
Plan to Share IPD: No